CLINICAL TRIAL: NCT01814345
Title: "An Observational Study to Determine the Incidence of of Her 2 Positivity in 100 Consecutive Gastric Cancers"
Brief Title: Her 2 Testing in Indian Patients With Gastric Cancer
Status: Terminated | Type: Observational
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Principal Investigator, Dr Bhawna Sirohi, Consulting Medical Oncologist, Tata Memorial Hospital
Other Study IDs: 1077; Her 2 in gastric cancer (Other Grant/Funding Number: Roche pharma limited)
Record Dates: First submitted 2013-02-27; First posted 2013-03-19 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Gastric Cancer
Keywords: Her2 testing (Human Epidermal Growth Factor Receptor 2)
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Gastric cancer remains a major health issue and a leading cause of cancer death worldwide, although the prevalence and mortality of the disease have gradually decreased. The investigators have very few options for patients with advanced disease.

The trastuzumab for Gastric Cancer (ToGA) trial, a pivotal randomized clinical trial of patients with HER-2 positive advanced, mostly metastatic, gastric cancer, proved the efficacy of trastuzumab (anti-Her 2 therapy) in combination with chemotherapy. The median overall survival was significantly prolonged in the trastuzumab-containing arm (13.8 vs. 11.1 months; HR 0.74; p=0.0046) without unexpected toxicity including cardiac events. The survival benefit was most pronounced in the subgroup of high HER-2/neu protein overexpression (median overall survival of 16 months). Only 20% of the patients screened and subsequently enrolled for this study were found to be HER2-positive when utilizing both immunohistochemistry and FISH. Her2 testing is recommended for all patients with advanced gastric cancers and type III oesophageal adenocarcinomas.

Data on Indian patients is lacking. Hence, the investigators plan to test for Her 2 in 100 patients with IHC and FISH in 2+ and 3+ patients.

DETAILED DESCRIPTION:
1. Study Objective/ Aims Aim: - Rate of Her 2 positivity in 100 consecutive gastric cancer patients Primary Objective

   Test for Her 2 in 100 consecutive gastric cancer patients Immuno-histochemistry will be done in all patients. Patients with 2 and 3+ IHC will also have FISH done.
2. Study Design& Methodology

   Patients will have the Her2 tested in 100 consecutive gastric cancer samples by immunohistochemistry and patients with 2+ and 3+ result will also have FISH done. This will not affect patient management
3. Overview of Data collection Dr.Bhawna Sirohi the principal investigators will maintain and supervise data collection and maintaining records. The patient will be de-identified.
4. Selection of Study Population

Inclusion Criteria:

100 consecutive patients with gastric cancer who have a pathology specimen at TMH

Exclusion Criteria:

If histopathology blocks were not available

5) Sample size 100 to be enrolled. Patient consent waiver applied for as this does not affect patient care 6) Statistical Analysis It is an Observational study so Results will be given as %age of total population.

ELIGIBILITY:
Inclusion Criteria:

* 100 consecutive patients with gastric cancer who have a pathology specimen at TMH

Exclusion Criteria:

* If histopathology blocks were not available

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 consecutive Gastric Cancer
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Incidence of Her2 testing in Gastric cancer | 6 month
  Immuno-histochemistry will be done in all patients. Patients with 2 and 3+ IHC will also have FISH done.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Bhawna Sirohi, MBBS DCH, Principal Investigator — Consulting Medical Oncologist; Shailesh Shrikhande, MS, Principal Investigator — Professor of Surgical GI and HPB surgery; Mukta Ramadwar, MD, Principal Investigator — Consultant Pathologist
Locations (1):
- Tata Memorial Hospital, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: Undecided